CLINICAL TRIAL: NCT06524427
Title: Robot-Assisted Versus Video-Assisted Lobectomy for Non-Small Cell Lung Cancer (RAVAR): A Multicenter, Open-Label, Randomized, Non-Inferiority Trial
Brief Title: Robot-Assisted vs. Video-Assisted Lobectomy for NSCLC (RAVAR)
Acronym: RAVAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Qingdao University (Other); The General Hospital of Eastern Theater Command (Other); Gansu Provincial Hospital (Other); Tang-Du Hospital (Other); Wuhan TongJi Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); West China Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shenzhen People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shandong Provincial Hospital (Other Government); Jiangsu Cancer Institute & Hospital (Other); Guangdong Provincial People's Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Qilu Hospital of Shandong University (Other); Jiangxi Provincial People's Hopital (Other); Sichuan Cancer Hospital and Research Institute (Other); Lanzhou University Second Hospital (Other); Shenzhen Third People's Hospital (Other); Qianfoshan Hospital (Other); Guangxi Nanxishan Hospital (Unknown)
Responsible Party: Principal Investigator, Hao-Xian Yang, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-5010-2019-04; ChiCTR2000034737 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2024-07-11; First posted 2024-07-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Robotic-assisted lobectomy; Video-assisted lobectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RATS group (Experimental): Patients will receive robot-assisted lobectomy
  Interventions: Procedure: Robot-assisted lobectomy
- VATS group (Active Comparator): Patients will receive video-assisted lobectomy
  Interventions: Procedure: Video-assisted lobectomy

INTERVENTIONS:
Procedure: Robot-assisted lobectomy — Patients will receive robot-assisted lobectomy using Da Vinci surgical system
  Arms: RATS group
Procedure: Video-assisted lobectomy — Patients will receive video-assisted lobectomy
  Arms: VATS group

SUMMARY:
Video-assisted thoracic surgery (VATS) has been recommended by clinical guidelines as one of the preferred surgeries for early-stage non-small cell lung cancer (NSCLC) for many years. However, VATS has inherent drawbacks, so at the beginning of this century, robotic-assisted thoracoscopic surgery (RATS) was first applied for lung resection. In recent years, RATS has developed rapidly, but there are still many unsolved scientific problems in the field of RATS. Thus, a multicenter prospective randomized controlled trial was conducted with stage I-II NSCLC patients as the study subject and 5-year DFS as the primary endpoint to compare the short-term and long-term outcomes of RATS and VATS in the treatment of early-stage NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years old;
2. Patients with blood pressure<160/100mmHg, 5.6<blood glucose<11.2mmol/L, major organs function normally: (1) Goldman index between grade 1 and 2; (2) Predicted forced expiratory volume in 1s (FEV1) >= 40 % and diffusing capacity of the lung for carbon monoxide (DLCO) >= 40 %; (3) total bilirubin <= 1.5 upper limit of normal; (4) Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) <= 2.5 upper limit of normal; (5) creatinine <= 1.25 upper limit of normal and creatinine clearance rate (CCr) >= 60ml/min;
3. The first clinical diagnosis before surgery was non-small cell lung cancer, including adenocarcinoma, squamous cell carcinoma, large cell carcinoma, and other unknown types;
4. Clinical stage T1-2N0-1 (cI-II): Maximum diameter of tumor <= 5cm and short diameter of mediastinal lymph node <= 1cm in thin layer CT;
5. Performance status of Eastern Cooperative Oncology Group (ECOG) 0-1;
6. All relevant examinations were completed within 28 days before the operation;
7. Patients who understand this study and have signed an approved Informed Consent.

Exclusion Criteria:

1. Patients with radiotherapy, chemotherapy, targeted therapy, or immunotherapy before surgery.
2. Patients with the previous history of other malignancies;
3. Patients with secondary primary cancer when enrolled;
4. Patients diagnosed as pure ground glass opacity (GGO) before surgery;
5. Patients diagnosed as mixed GGO whose solid part <= 50% and Maximum diameter of tumor <= 2cm;
6. Patients with small cell lung cancer;
7. Patients with prior unilateral open thoracic surgical procedures;
8. Woman who is pregnant or breastfeeding;
9. Patients with interstitial pneumonia, pulmonary fibrosis, or severe emphysema;
10. Patients with an active bacterial or fungal infection that is difficult to control;
11. Patients with serious psychosis;
12. Patients with a history of severe heart attack, heart failure, myocardial infarction, or angina within the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1124 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival (DFS) | 5 years after surgery
  Difference of 5-year disease free survival rate between the two groups

SECONDARY OUTCOMES:
5-year overall survival (OS) | 5 years after surgery
  Difference of 5-year overall survival rate between the two groups
3-year disease-free survival (DFS) | 3 years after surgery
  Difference of 3-year disease free survival rate between the two groups
3-year overall survival (OS) | 3 years after surgery
  Difference of 3-year overall survival rate between the two groups
Blood loss | During the surgery
  Blood loss during the surgery
Conversion rate | During the surgery
  The number of patients converted to thoracotomy divided by the total number of included patients in a group
Perioperative complication | The day of surgery, 2/4/8/12/26/52 weeks after surgery
  Intraoperative and postoperative complications
Operative death rate | 30/90 days after surgery
  The number of patients died within 30/90 days after surgery divided by the total number of included patients in a group
Hospital stays after surgery | Between the date of surgery and the date of discharge, assessed up to 30 days
  The length of stay in hospital after surgery
Pain score after surgery | Scores were given daily after surgery and at weeks 2/4/8/12/26/52 after discharge
  The degree of pain after surgery was measured using Numerical Rating Scale (NRS). The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable). The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours.
R0 rate | Postoperative in-hospital stay up to 30 days
  The number of patients received R0 surgery divided by the total number of included patients in a group
Operative time | During the surgery
  The total time from skin to skin and the time of each step were recorded
The number of resected lymph nodes | Postoperative in-hospital stay up to 30 days
  The number of resected lymph nodes were calculated according to the official pathological report after surgery
Chest tube duration | Postoperative in-hospital stay up to 30 days
  The number of days between the date of surgery and the date of chest tube removal
Acesodyne (Grade III) dose | Postoperative in-hospital stay up to 30 days
  The total amount of morphine used by the patient during the postoperative hospital stay, including morphine, pethidine, and fentanyl etc.
Total cost of hospitalization | From the date of admission to the date of discharge, assessed up to 30 days
  The total cost of the patient from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Xian Yang, M.D., Principal Investigator — Sun Yat-sen University
Locations (23):
- China (23):
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Guangxi Nanxishan Hospital, Guilin, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan TongJi Hospital, Wuhan, Hubei
  - The General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hopital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - Tang-Du Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qianfoshan Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This clinical trial has been registered in Chinese Clinical Trial Registry with a registration number as ChiCTR2000034737 — https://www.chictr.org.cn/bin/project/edit?pid=48784